CLINICAL TRIAL: NCT00845767
Title: The Cardiovascular Effects of Air Pollution: the Role of Nitric Oxide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Umeå University (Other)
Responsible Party: Dr Jeremy P Langrish, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DNR 08-185M/1
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Endothelial Dysfunction
Keywords: Nitric Oxide; Nitric Oxide Synthase; Air Pollution; Endothelial Dysfunction; Diesel Exhaust

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diesel Exposure (Experimental): 1 hour exposure to dilute diesel exhaust at a concentration of 300 µg/m3 with intermittent exercise
  Interventions: Procedure: Forearm Vascular Study
- Air Exposure (Experimental): 1 hour exposure to filtered air during intermittent exercise
  Interventions: Procedure: Forearm Vascular Study

INTERVENTIONS:
Procedure: Forearm Vascular Study — Forearm venous occlusion plethysmography during intraarterial infusion of L-NMMA (2-8 µmol/min) followed by co-infusion of sodium nitroprusside (90-900 ng/min) as a "nitric oxide clamp". Forearm blood flow then measured during the clamp in response to infused vasodilators acetylcholine (5-20 mg/min), bradykinin (100-1000 pmol/min), verapamil (10-100 µg/min) and sodium nitroprusside (2-8 µg/min).
  Other Names: ACh; SNP; BK

SUMMARY:
Exposure to air pollution has been linked to increased cardiorespiratory morbidity and mortality. The exact component of air pollution that mediates this effect is unknown, but the link is strongest for fine combustion derived particulate matter derived from traffic sources. Recently, it has been demonstrated that inhalation of diesel exhaust impairs vascular vasomotor tone and endogenous fibrinolysis. The mechanism underlying these detrimental vascular is unclear, but is thought to be via oxidative stress and altered bioavailability of endogenous nitric oxide. In these studies we plan to elucidate the role of endogenous nitric oxide (NO) in the adverse vascular responses observed following exposure to diesel exhaust.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Use of regular medication (except oral contraceptive pill)
* Current smokers
* Significant occupational exposure to air pollution
* Intercurrent illness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow as measured by venous occlusion plethysmography during infusion of NOS inhibitors and vasodilators | 2-4 hours after exposure

SECONDARY OUTCOMES:
Plasma nitrite concentrations | During forearm study
Plasma concentrations of t-PA and PAI | After infusion of bradykinin during forearm study

CONTACTS AND LOCATIONS:
Overall Officials: Anders Blomberg, MD PhD, Principal Investigator — Umeå University; David E Newby, PhD FRCP, Principal Investigator — University of Edinburgh
Locations (1):
- Umeå University, Umeå, Sweden

REFERENCES:
- [Background] Mills NL, Tornqvist H, Robinson SD, Gonzalez M, Darnley K, MacNee W, Boon NA, Donaldson K, Blomberg A, Sandstrom T, Newby DE. Diesel exhaust inhalation causes vascular dysfunction and impaired endogenous fibrinolysis. Circulation. 2005 Dec 20;112(25):3930-6. doi: 10.1161/CIRCULATIONAHA.105.588962. PMID 16365212
- [Derived] Langrish JP, Unosson J, Bosson J, Barath S, Muala A, Blackwell S, Soderberg S, Pourazar J, Megson IL, Treweeke A, Sandstrom T, Newby DE, Blomberg A, Mills NL. Altered nitric oxide bioavailability contributes to diesel exhaust inhalation-induced cardiovascular dysfunction in man. J Am Heart Assoc. 2013 Feb 19;2(1):e004309. doi: 10.1161/JAHA.112.004309. PMID 23525434